CLINICAL TRIAL: NCT07183696
Title: Effect of Breath Booster Training on Respiratory Muscle Strength and Quality of Life in Hemodialysis Patients
Brief Title: Respiratory Muscle Training and Quality of Life in Hemodialysis Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sameh Eldaly, director of scientific research committee, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/005826
Record Dates: First submitted 2025-09-11; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Hemodialysis
MeSH Terms: interventions — Breathing Exercises; Vibration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): will receive respiratory physical therapy sessions in the form of breathing exercises, chest percussion, and vibration 3 times per week during dialysis sessions for 6 weeks
  Interventions: Other: breathing exercises
- Intervention Group (Experimental): will receive respiratory physicaltherapy sessions in the form of breathing exercises, chest percussion, and vibration 3 times per week during dialysis sessions for 6 weeks and training on the breath booster device at the same session
  Interventions: Other: breathing exercises

INTERVENTIONS:
Other: breathing exercises — * breathing exercises as needed 3 times per week during dialysis sessions.
  * chest percussion as needed 3 times per week during dialysis sessions.
  * vibration as needed 3 times per week during dialysis sessions.
  Other Names: chest percussion; vibration

SUMMARY:
This study investigates the effect of breath booster training on respiratory muscle strength and quality of life in patients undergoing hemodialysis. It aims to determine whether targeted respiratory training can improve pulmonary function, enhance physical performance, and positively impact overall well-being in this population.

DETAILED DESCRIPTION:
Detailed Description Statement of the problem Does Breath Booster training have an effect on respiratory muscle strength and quality of life in hemodialysis patients? Purpose of the study

The study aims to:

Investigate the effect of the Breath Booster device on respiratory muscle strength in patients undergoing dialysis.

Evaluate the impact of the Breath Booster device on the quality of life of patients undergoing dialysis.

Assess the effect of the Breath Booster device on exercise capacity in dialysis patients.

Significance of the study The burden of chronic kidney disease (CKD) in Egypt has increased significantly over the past decade, with a 36% rise in cases between 2009 and 2019. CKD is now the fifth leading cause of death in the country, highlighting the urgent need for effective patient-centered interventions. A 2024 report underscored the importance of implementing a comprehensive renal registry to improve patient outcomes and lessen the healthcare burden.

Hemodialysis patients face substantial challenges, including adherence to strict dietary and fluid restrictions, repeated dialysis sessions each week, and vascular access care. These lifestyle demands often contribute to reduced physical function, lower quality of life, and increased psychological stress.

Moreover, respiratory muscle weakness is a common complication among CKD patients, particularly those on hemodialysis. This impairment reduces functional capacity and negatively impacts quality of life. Inspiratory muscle training (IMT) has recently emerged as a promising, non-pharmacological method to address this issue.

Given these factors, the present study seeks to evaluate the effectiveness of the Breath Booster device in improving respiratory muscle strength, quality of life, and exercise capacity in hemodialysis patients.

Delimitation

This study will be delimited to:

Forty patients participating in the study. Age range between 50-60 years. Patients diagnosed with end-stage renal disease (CKD stage 5) on hemodialysis. Patients who have been undergoing regular hemodialysis for 1-3 years.

Null Hypothesis There will be no significant effect of Breath Booster training on respiratory muscle strength and quality of life in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

1. Fifty patients will be included in this study.
2. Their ages will range from 50 to 60 years.
3. Patients with end-stage renal disease (grade 5) receiving hemodialysis.
4. Patients on hemodialysis for around 1 to 3 years.
5. They will be able to follow instructions during evaluation and treatment.

Exclusion Criteria:

1. Diabetes Mellitus,
2. Morbid obesity with a BMI of more than 35 kg/m2.
3. Hearing or visual impairments.
4. Any severe chest diseases like COPD.
5. Certain contraindications for the use of the Breath Booster. Individuals with severe respiratory conditions such as unstable asthma, or emphysema, or those who have recently undergone lung surgery
6. Uncontrolled seizures.

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Respiratory Muscle Strength measured using Respiratory Pressure Manometers | 6 weeks
  Outcomes include maximum inspiratory pressure (MIP) and maximum expiratory pressure (MEP), recorded in cmH₂O. Higher values indicate greater respiratory muscle strength.
Health-Related Quality of Life assessed by the 36-Item Short Form Health Survey | for 6 weeks
  It includes eight domains (physical functioning, role limitations, bodily pain, general health, vitality, social functioning, role-emotional, and mental health). Scores are transformed to a 0-100 scale, where 0 = worst health and 100 = best health. Higher scores indicate better health-related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No